CLINICAL TRIAL: NCT03035123
Title: Impact of an Intensive Therapeutic Education on Occurrence of Clinical Events in Patients With Acute Heart Failure: EduStra-HF Study
Brief Title: Therapeutic Education Strategy for Patients With Acute Heart Failure
Acronym: EduStra-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Resicard (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government); Assistance Publique - Hôpitaux de Paris (Other); French Cardiology Society (Other)
Responsible Party: Principal Investigator, Pr Ariel Cohen, Head of the cardiology department, Saint Antoine University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EduStra-HF; RCB ID: 2016-A00899-42 (Other Grant/Funding Number: National Drug and Health Products Safety Agency (ANSM))
Record Dates: First submitted 2016-12-05; First posted 2017-01-27 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Heart Failure; Therapeutic education; Quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Usual care" (No Intervention): Patients will attend an appointment with the therapeutic education nurse before discharge, after which they will have no further contact with the education team. The Research team members will telephone the patient three times during the year (after 2, 6 and 12 months) to collect data on HF treatments, blood tests results, health-related events and hospitalizations.
- Interventional (Experimental): Before discharge, patients will attend an appointment with a nurse trained in therapeutic education, in which the nurse will evaluate the overall knowledge and the skills of the patient about HF. The nurse will then define specific educational objectives with the patient, based on the patient's medical history, state of disease, comorbidities, alarm signs, fears and knowledge.
  Each patient will receive six telephone calls and two home-visits during the 1 year of follow-up. Each contact between the nurse and the patient will be dedicated to HF education. The patient will also receive regular short text messages containing health advice and appointment reminders.
  To help the patient regain his/her autonomy, intervals between education sessions will be progressively longer.
  Interventions: Behavioral: Therapeutic education

INTERVENTIONS:
Behavioral: Therapeutic education — Interventional arm
  Arms: Interventional

SUMMARY:
The EduStra-HF study will examine the impact of an intensive therapeutic education on patients discharged from hospital after an episode of acute heart failure (HF).

Patients will be randomized into two groups: one will receive "usual care" monitoring and one will receive a specific educational monitoring programme for 1 year.

All patients will meet with a specialized therapeutic education nurse before discharge.

The effect of the intensive education on HF rehospitalization and quality of life will be examined.

DETAILED DESCRIPTION:
The prevalence of HF in France is increasing. According to a report from the Haute Autorité de Santé (HAS) - the French Health Authority - published in June 2015 concerning discharge of patients hospitalized for HF, 2.3% of the French adult population is affected. Despite improvements in treatment and HF-specific care, the rehospitalization rate for HF remains substantial, and HF management is a major public health issue.

Chronic HF leads to psychological and physiological issues in patients. Furthermore, this disease affects patient quality of life and activities of daily living.

The HAS also reported that even if iterative hospitalizations are the consequence of complicated and multifactorial situations, some could be prevented by improved patient care.

The aim of the EduStra-HF study is to examine the effect of an intensive therapeutic education on patients discharged from hospital after an episode of acute HF. It will study whether this intervention reduces the rate of rehospitalization and increases quality of life in this population.

To achieve this goal, a multicentre, randomized, two parallel arm study will be conducted. Patients will be included in several cardiology centres in Paris (Ile-de-France) over 2 years and 3 months.

Included patients, chosen from patients admitted for acute HF in the participating hospitals, will be randomized into two groups, which will determine the monitoring they receive after discharge. For each patient, monitoring will last for 1 year from the day they return home.

The first group of patients will be randomized to receive "usual care" monitoring and will not be given specific therapeutic education after discharge.

The second group (intervention arm) will receive a specific educational monitoring programme from nurses via telephone calls and home visits, for 1 year. Monitoring will began early after discharge. Annual medical monitoring and visits to the cardiologist will also be planned.

All patients, regardless of attribution arm, will meet a nurse trained in therapeutic education during their stay in hospital. Moreover, validated and HF-related self-assessed questionnaires will be analyzed to assess quality of life and impact of HF on patient activities of daily living.

In the interventional arm, patients will receive monitoring documents, such as a HF information booklet and a personal monitoring agenda.

The EduStra-HF study will provide a specific analysis of a multisupport therapeutic education (including medical monitoring). Data on all HF drug treatments, including the more recent ones (e.g. Entresto), blood tests results, and cardiologic data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with acute HF
* Affiliated to the French Social Security system
* Accepting the principle of telephone monitoring
* Accepting home visits from a study nurse
* Possession of a mobile phone

Exclusion Criteria:

Psychosocial:

* Refusal to accept the study design
* Patient under guardianship
* Monitoring obstacle: language, cognitive deficiency, itinerant lifestyle, regular travel, institutionalization
* Inability to sign the consent form or to complete questionnaires

Medical:

* Active cancer
* Severe psychiatric or neurological disorder
* Complicated acute myocardial infarction
* Significant valvular diseases requiring surgery
* Hypertrophic obstructive cardiomyopathy
* Planned heart transplant
* Cardiac surgery in the previous 3 months
* Enrollment in another clinical trial
* Medical or surgical procedure which might interfere with monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Number of rehospitalizations for acute heart failure (HF) in both groups of patients | 1 year

SECONDARY OUTCOMES:
Patients knowledge about the illness | 1 year
  Nurses will evaluate during each telephone call and home visit patients knowledge and skills about the following items : illness, treatments, diet, physical activity, medical follow-up. This data will be recorded in a specific table and classified into "acquired / partially acquired / not acquired" items.
Global quality of life | 1 year
  Assessed by validated questionnaire SF-12
Quality of life linked to Heart Failure | 1 year
  Assessed by validated questionnaire KCCQ-15
Length of stay for HF and all-cause hospitalizations | 1 year of follow-up
Hospitalization rate for cardiovascular diseases except HF | 1 year of follow-up
Cardiovascular and all-cause mortality rate | 1 year of follow-up
B-type natriuretic peptide (BNP) or NT pro-BNP levels | During 1 year of follow-up

OTHER OUTCOMES:
Cost effectiveness of the intervention | During 1 year of follow-up
  Comparison between both groups of patients of the HF-hospitalizations average cost, related to the operating cost of the EduStra-HF method.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Cohen, MD PhD, Principal Investigator — Hôpital Saint-Antoine
Locations (6):
- France (6):
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Clinique du Mont Louis, Paris
  - Hopital AP-HP Saint-Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Cardiologique du Nord, Saint-Denis
  - Centre Hospitalier André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: Undecided
Sharing Individual Participant Data requires a specific authorization from the French Board CNIL (Commission Nationale de l'Informatique et des Libertés) which chooses whether to allow the research team to share patient data. A specific request is needed and will be sent to that authority.

REFERENCES:
- [Derived] Jullien S, Lang S, Gerard M, Soulat-Dufour L, Brito E, Ocokoljic E, Laperche T, Georges JL, Diakov C, Belliard O, Larrazet F, Bataille S, Assyag P, Cohen A; EduStra-HF investigators. Intensive therapeutic education strategy for patients with acute heart failure (EduStra-HF): Design of a randomized controlled trial. Arch Cardiovasc Dis. 2024 Oct;117(10):561-568. doi: 10.1016/j.acvd.2024.04.006. Epub 2024 Jul 4. PMID 39089896